CLINICAL TRIAL: NCT02723136
Title: Implementing a Smartphone Application to Optimise Academic Performance Among Medical Students: A Randomised Trial
Brief Title: Implementation of a Smartphone Application in Medical Education
Acronym: iSTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Laboratorio de Ingeniería y Tecnología (LABITEC) (Unknown)
Responsible Party: Principal Investigator, Felipe Martinez, Professor, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CEC098-16
Record Dates: First submitted 2016-03-27; First posted 2016-03-30 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Education, Medical
Keywords: Smartphone; Internship; Internal Medicine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone application (Experimental): Participants allocated to this arm will receive a smartphone application developed to assist and guide the study of internal medicine and its subspecialties. The application will provide feedback to participants regarding their overall performance in terms of correct answers and the overall time required to solve a clinical vignette.
  Interventions: Device: Smartphone Application
- Usual care (No Intervention): Students allocated to this arm will not receive any further assistance in studying for this trial's tests.

INTERVENTIONS:
Device: Smartphone Application — Smartphone application developed by internists and engineers. Will be made available on iOS(R) and Android(R) operating systems.
  Arms: Smartphone application

SUMMARY:
This study addresses the effectiveness of a smartphone application to improve academic performance among medical students. Participants will be randomised to receive an application developed by a team of physicians and engineers, designed to review key concepts in internal medicine and its subspecialties. The primary outcome will be the number of correct answers in a multiple choice test 4 weeks after randomisation.

DETAILED DESCRIPTION:
Smartphones are devices that are commonly used by medical professionals. Their adoption by students and physicians is increasing, with reported use rates of roughly 85%. Reasons behind these implementation rates stem from their versatility, since this technology provides mobile communications and advanced informatics in a handheld device that can be used at the bedside. However, data regarding their use in medical education is scarce.

This study aims to address whether a smartphone application designed to review key concepts in internal medicine and its subspecialties might increase the overall academic performance of medical students. Eligible participants will be interns in their final year of study who own a smartphone with an operating system based in Android® or iOS®. Only those that do not wish to participate will be excluded from this trial.

All participants will undergo a baseline test aimed at addressing their knowledge of internal medicine and its subspecialties. Multiple choice questions will be used in this test, which have been developed by a team of internists with 5 years experience in formulating them. These questions have also been designed to resemble a national examination that is required to practice medicine in the Chilean Public Health System, and have shown a good correlation with performance in the latter exam in previous reports. In order to optimise adherence, the application will also provide feedback to its user, showing overall performance in terms of correct answers and time required to solve a clinical vignette.

After this test, participants will be randomised to receive the smartphone application by a statistician. Investigators will be kept unaware of the allocation sequence used in this trial. The contents of the application will include clinical vignettes that will review core concepts in internal medicine and its subspecialties. After 4 weeks, participants will undergo a second test and the overall performance between groups will be compared. Both outcome assessors and statisticians will be kept unaware of participant allocation. Data regarding the overall application use will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* Medical student coursing their internship.
* Owns a smartphone with an Android® or iOs®-based operating system

Exclusion Criteria:

* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Academic Performance | 4 weeks after randomisation
  Overall percentage of correct responses in a standardised test.

SECONDARY OUTCOMES:
Time to complete tests | 4 weeks after randomisation
  Time required by students to complete a 90-question multiple-choice test.

OTHER OUTCOMES:
Application adherence | 4 weeks after randomisation
  Mean time spent using the application.
Application adherence | 4 weeks after randomisation
  Mean number of questions answered by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Martinez, M.D., M.Sc., Principal Investigator — Universidad de Valparaiso
Locations (1):
- Campus de la Salud, Universidad de Valparaiso, Reñaca, Viña Del Mar, Chile

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make individual participant data available.

REFERENCES:
- [Background] Mosa AS, Yoo I, Sheets L. A systematic review of healthcare applications for smartphones. BMC Med Inform Decis Mak. 2012 Jul 10;12:67. doi: 10.1186/1472-6947-12-67. PMID 22781312
- [Background] Shah J, Haq U, Bashir A, Shah SA. Awareness of academic use of smartphones and medical apps among medical students in a private medical college? J Pak Med Assoc. 2016 Feb;66(2):184-6. PMID 26819165
- [Background] Baumgart DC. Smartphones in clinical practice, medical education, and research. Arch Intern Med. 2011 Jul 25;171(14):1294-6. doi: 10.1001/archinternmed.2011.320. No abstract available. PMID 21788549
- [Background] Rung A, Warnke F, Mattheos N. Investigating the use of smartphones for learning purposes by Australian dental students. JMIR Mhealth Uhealth. 2014 Apr 30;2(2):e20. doi: 10.2196/mhealth.3120. PMID 25099261
- [Background] O'Connor P, Byrne D, Butt M, Offiah G, Lydon S, Mc Inerney K, Stewart B, Kerin MJ. Interns and their smartphones: use for clinical practice. Postgrad Med J. 2014 Feb;90(1060):75-9. doi: 10.1136/postgradmedj-2013-131930. Epub 2013 Nov 15. PMID 24243966
- See also: National Examination that enables physicians to practice medicine in the public health system — http://www.eunacom.cl/